CLINICAL TRIAL: NCT05098730
Title: Strategy Training and Pets to Promote Stroke Survivor's Cognitive Performance and Community Participation
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Haifa (Other)
Responsible Party: Principal Investigator, Naor Demeter, Principal Investigator, Faculty Associate, University of Haifa
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: STUDY21080031
Record Dates: First submitted 2021-10-15; First posted 2021-10-28 (Actual); Last update posted 2024-08-09 (Actual); Status verified 2024-08

CONDITIONS: Stroke
MeSH Terms: conditions — Stroke

STUDY DESIGN:
Intervention Model Description: The proposed study is a single site, two-group quasi-experimental design comparing the effects of strategy training on rehabilitation engagement, cognitive performance, and community participation of home-dwelling stroke survivors living with and without pets. The investigators will also conduct qualitative interviews with participants who have pets.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Stroke survivors with pets (Experimental): Stroke survivors with pets will receive strategy training for 10-15 sessions, 45 minutes each session, delivered by a trained occupational therapist in the home.
  Interventions: Behavioral: Strategy Training
- Stroke survivors without pets (Active Comparator): Stroke survivors without pets will receive strategy training for 10-15 sessions, 45 minutes each session, delivered by a trained occupational therapist in the home.
  Interventions: Behavioral: Strategy Training

INTERVENTIONS:
Behavioral: Strategy Training — Strategy training is comprised of participant-selected activity based goals, self evaluation, global problem solving strategies, and therapist-delivered guided training. The strategy training therapist will guide participants using prompting questions, as well as work sheets that facilitate learning and aid the participants in implementing the process.

SUMMARY:
The study will administer an intervention called strategy training to adult stroke survivors living in the community who do and do not have pets, and will examine the role of a pet in promoting cognitive performance and community participation outcomes.

ELIGIBILITY:
Stroke survivors with pets

Inclusion Criteria:

1. Primary diagnosis of acute stroke
2. At least 3 months after the stroke onset
3. Living in a community residence with a pet
4. Cognitive impairment as indicated by an Executive Interview score of 3 or higher
5. Participation restrictions as indicated by an Activity Card Sort (<80% of pre-stroke activities)
6. Willing to participate in a 6-week program with 2 intervention sessions per week at home

Exclusion Criteria:

1. Dementia as indicated by Montreal Cognitive Assessment score of 18 or lower
2. Severe aphasia as indicated by the Boston Diagnostic Aphasia Examination Severity Score of 0 or 1
3. Self-report of a central nervous system disorder other than stroke
4. Recent drug or alcohol addiction/abuse within 3 months prior to the Mini-Neuropsychiatric Interview
5. Severe mental illness as indicated by the PRIME-MD
6. Prior exposure to strategy training
7. Currently participate in rehabilitation therapy programs

Stroke survivors without pets

Inclusion Criteria:

1. Primary diagnosis of acute stroke
2. At least 3 months after the stroke onset
3. Living in a community residence
4. Cognitive impairment as indicated by an Executive Interview score of 3 or higher
5. Participation restrictions as indicated by an Activity Card Sort (<80% of pre-stroke activities)
6. Willing to participate in a 6-week program with 2 intervention sessions per week at home

Exclusion Criteria:

1. Dementia as indicated by Montreal Cognitive Assessment score of 18 or lower
2. Severe aphasia as indicated by the Boston Diagnostic Aphasia Examination Severity Score of 0 or 1
3. Self-report of a central nervous system disorder other than stroke
4. Recent drug or alcohol addiction/abuse within 3 months prior to the Mini-Neuropsychiatric Interview
5. Severe mental illness as indicated by the PRIME-MD
6. Prior exposure to strategy training
7. Currently participate in rehabilitation therapy programs

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2024-10-01 (Estimated); Primary Completion 2025-12-31 (Estimated); Study Completion 2026-06-30 (Estimated)

PRIMARY OUTCOMES:
Mean engagement score as measured by the Pittsburgh Rehabilitation Participation Scale | Baseline to 6 weeks
  The scale is a valid and reliable criterion referenced measure that assesses engagement in rehabilitation therapy sessions. Each session is scored by the occupational therapist, 1 (no participation, refusal) to 6 (excellent participation). Scores are averaged across the 10-15 intervention sessions to generate the mean engagement score.

SECONDARY OUTCOMES:
Change in attention as measured by the Color Trail Test 1 | Baseline to 3 months
  This measure assesses perceptual tracking, sustained attention and grapho-motor skills. It is a pencil and paper, timed test. Completion time in seconds for each task is recorded, with a lower score representing better function. Change in attention will be calculated by subtracting the time to do the task at baseline from the time to do the task at 3 months.
Change in executive function as measured by the Color Trail Test 2 | Baseline to 3 months
  This measure assesses divided attention and sequencing skills, which are executive function performance. It is a pencil and paper, timed test of effortful executive processing abilities that assesses the ability to alternate between two colors. Completion time in seconds for each task is recorded, with a lower score representing better function. Change in executive function will be calculated by subtracting the time to do the task at baseline from the time to do the task at 3 months.
Change in community participation as measure by Community Participation Indicators score | Baseline to 3 months
  This participant reported questionnaire will measure the frequency of community participation over a 7 days period. Each item is measured on a 5-point Likert scale, with 1=no participation in that activity and 5=7 days of participation in that activity. A total of 20 items are summed to yield a total score. Change in community participation will be calculated by subtracting baseline total score from the 3 month total score.

CONTACTS AND LOCATIONS:
Overall Officials: Naor Domotor, PhD, Principal Investigator — University of Pittsburgh
Locations (1):
- University of Pittsburgh, Pittsburgh, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: No